CLINICAL TRIAL: NCT06767722
Title: Effectiveness of a Lifestyle Intervention for Pregnant Women With Abnormal Glucose Metabolism in Early Pregnancy: EAGM Randomized Controlled Trial
Brief Title: Effectiveness of a Lifestyle Intervention for Pregnant Women With Abnormal Glucose Metabolism in Early Pregnancy: EAGM Trial
Acronym: EAGM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Jiangmen Maternity and Child Health Care Hospital (Unknown); Panyu Maternal And Child Care Service Centre Of Guangzhou (Unknown); The Affiliated Shunde Hospital of Jinan University (Unknown); Shenzhen Second People's Hospital (Other); Guangxi Hospital Division of The First Affiliated Hospital, Sun Yat-sen University (Unknown); BoAi Hospital of Zhongshan (Other); Yuebei People's Hospital (Other); Qingyuan People's Hospital (Other); The Sixth Affliated Hospital of Jinan University (Unknown); Baoan Maternal And Child Health Care Hospital, Shenzhen, China (Unknown); Jiangxi Maternal and Child Health Hospital (Other); Guangxi provincial maternal and chidren's hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Obstetrics and Gynecology Hospital of Zhejiang University (Unknown); Xiangya Hospital of Central South University (Other); Guangzhou Women's and Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Haitian Chen, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: [2024]645
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Early Pregnancy; Fasting Plasma Glucose; Hemoglobin A1c Protein, Human; Lifestyle Intervention; Adverse Pregnancy Outcomes
MeSH Terms: interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The Intervention group will receive both intervention and routine prenatal care.
  Interventions: Behavioral: Lifestyle intervention and self-monitoring of blood glucose
- control group (No Intervention): The control group will only receive routine prenatal care.

INTERVENTIONS:
Behavioral: Lifestyle intervention and self-monitoring of blood glucose — The intervention will consist of a lifestyle intervention that comprises advice on diet, exercise, weight management, and self-monitoring of blood glucose (SMBG) with feedback from healthcare professionals on results and insulin treatment if indicated.
  Arms: intervention group

SUMMARY:
This is a multicentre, parallel-group, open-label, pragmatic, randomised-control trial of early lifestyle intervention versus routine prenatal care by random allocation (1:1) in women with early abnormal glucose metabolism (EAGM) to compare the incidence of large-gestational age and preterm birth between two groups. The investigators aim to assess the effectiveness of early lifestyle interventions and to provide evidence for the optimal standard management for Chinese women with EAGM.

DETAILED DESCRIPTION:
Women with early abnormal glucose metabolism (EAGM) , which is defined as fasting plasma glucose (FPG) 5.1-6.9 mmol/L and/or hemoglobin A1c (HbA1c) 5.7%-6.4% at before 14 weeks of gestation, will be recruited and randomized in a 1:1 ratio into the intervention or control group. The intervention will consist of a lifestyle intervention that comprises advice on diet, exercise, weight management and self-monitoring of blood glucose (SMBG) with feedback from healthcare professionals on results and insulin treatment if indicated. The educational session is delivered as an initial session following randomization followed by five follow-up sessions which will occur approximately every four months, either face-to-face during routine prenatal visits or via telephone consultation. Routine prenatal care will also be applied to the intervention group. Women in the control group will only receive routine prenatal care. Both groups will receive an OGTT test at 24-28 weeks of gestation unless insulin is needed before the OGTT test for suboptimally controlled blood glucose levels. Whether to continue the intervention depends on the OGTT results as women diagnosed with GDM or overt diabetes will continue intervention plus routine prenatal care until delivery while those will normal OGTT result will pause interventions and follow the routine prenatal care only until delivery. The primary outcome of our trial will be a composite of neonatal outcome including large-for-gestational age and preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Able to provide informed consent.
* Confirmed viable pregnancy on a nuchal translucency scan done between 11+0 and 13+6 weeks.
* Singleton pregnancies.
* An abnormal glucose metabolism determined by a blood test performed before 14 weeks, defined as FPG 5.1-6.9mmol/L and/or HbA1c 5.7-6.4%.

Exclusion Criteria:

* Pregestational diabetes (diagnosed as diabetes mellitus before pregnancy, or FPG≥7.0mmol/L, or HbA1c≥6.5% at the first prenatal visit), impaired fasting glucose or impaired glucose tolerance diagnosed before pregnancy.
* Plan for termination of pregnancy due to fetal anomaly identified at the first trimester scan.
* Use of medications known to interfere with glucose metabolism (e.g. corticosteroids, antipsychotic drugs) at the time of randomisation.
* Any other physical (serious medical conditions such as cancer, organ failure, epilepsy, paraplegia, disability) or psychological condition (e.g. learning difficulties, serious mental illness) that is likely to interfere with the conduct of the trial according to evaluation by the trial monitoring group.
* Women currently with hyperemesis gravidarum leading to dehydration or requiring hospitalization. If persisting vomiting resolves, the patient may be reassessed for inclusion in the trial up to and including 14+6 weeks of gestation, providing all other inclusion and exclusion criteria are met.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3430 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite neonatal outcome of large-gestational age and preterm birth | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.

SECONDARY OUTCOMES:
Pregnancy-related hypertensive disorders | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Gestational diabetes mellitus | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Gestational hypertension | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Preeclampsia | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Eclampsia | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Prescription of hypoglycaemic drug | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Preeclampsia requiring delivery before 37 weeks | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Total gestational weight gain | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Mode of birth | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Primary caesarean | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Large-for-gestational age | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Preterm birth at <37 weeks of gestation | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Neonatal birthweight | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Small-for-gestational-age | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Gestational age at birth, weeks and days | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Neonatal hypoglycaemia | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Admission to neonatal wards or intensive care unit | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Fetal loss <24 weeks of gestation | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Fetal loss ≥24 weeks of gestation | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Termination of pregnancy | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Neonatal death | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Apgar score at 1min after birth | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.
Apgar score at 5min after birth | outcomes will be collected up to primary hospital discharge, or 28 days after the estimated date of delivery, whichever is sooner.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yatsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes